CLINICAL TRIAL: NCT06236789
Title: Observation Study to Evaluate the Efficacy and Safety of Ifosfamide/Mesna in Patients With Metastatic Castration-resistant Prostate Cancer
Status: Recruiting | Type: Observational
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Other Study IDs: 4-2023-1306
Record Dates: First submitted 2024-01-24; First posted 2024-02-01 (Actual); Last update posted 2024-02-01 (Actual); Status verified 2024-01

CONDITIONS: Prostatic Neoplasm
Keywords: Castration-resistant prostate cancer; Ifosfamide/mesna; Efficacy; Safety
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Ifosfamide; Mesna

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Castration-resistant prostate cancer patients treated with ifosfamide/mesna
  Interventions: Drug: Ifosfamide/mesna

INTERVENTIONS:
Drug: Ifosfamide/mesna — Ifosfamide 2,500 mg/m2/day for 3 days every 3 weeks with mesna until disease progression

SUMMARY:
Prostate cancer is the 2nd most common cancer in men worldwide. Based on the results of several recent clinical trials, systemic treatments including hormone inhibitors, docetaxel, cabazitaxel, and PARP inhibitors are being used as standard treatment for patients with metastatic castration-resistant prostate cancer. However, there is insufficient research on salvage therapy for patients with metastatic castration-resistant prostate cancer who have failed standard treatment. In this study, the investigators will evaluate the effectiveness and safety of ifosfamide in castration-resistant prostate cancer by analyzing the treatment outcomes of patients who received ifosfamide/mesna treatment as salvage therapy.

DETAILED DESCRIPTION:
1. Retrospective analysis of the treatment outcomes of patients with metastatic castration-resistant prostate cancer who who received ifosfamide/mesna will be conducted.
2. Information regarding demographics (age, gender, and etc.), disease status (stage, metastatic lesion, and etc.), treatment details (administered anticancer drugs, treatment response to drug, and disease progression with progression date), and survival (death with date of death) will be recorded.
3. Statistical method was applied to analyze the correlation between clinical indicators and survival rate.

ELIGIBILITY:
Inclusion Criteria:

1. 19 years and older adult male
2. Patients with histologically confirmed prostate cancer
3. Castration-resistant prostate cancer
4. ECOG 2 or less
5. Patients with previous docetaxel exposure
6. Patients with available PSA level
7. Patients with evaluable disease based on RECIST 1.1

Exclusion Criteria:

1. Patients with other primary cancers diagnosed within 3 years other than prostate cancer
2. Patients with a history of organ transplantation
3. Hormone sensitive prostate cancer
4. ECOG 3 or higher
5. Patients without previous docetaxel exposure
6. Patients previously exposed to ifosfamide
7. Patients without available PSA level
8. Patients without evaluable disease based on RECIST 1.1

Min Age: 19 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Patients with prostate cancer
Study Population: Patients with metastatic castration-resistant prostate cancer
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2016-11 (Actual); Primary Completion 2026-11 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Objective response rate | Up to 2 years
  Summation of complete response partial response based on RECIST version 1.1

SECONDARY OUTCOMES:
Number of patients with Adverse events based on CTCAE | Up to 2 years
  Adverse events based on CTCAE
Overall survival | Up to 2 years
  From date of treatment start to death

CONTACTS AND LOCATIONS:
Overall Officials: Sang Joon Shin, Principal Investigator — Division of Medical Oncology, Department of Internal Medicine, Yonsei Cancer Center, Yonsei University College of Medicine
Locations (1):
- Division of Medical Oncology, Department of Internal Medicine, Yonsei Cancer Center, Yonsei University College of Medicine, Seoul, Republic of Korea, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided
Additional information reported in this study will be available upon request.

REFERENCES:
- [Derived] Kim CG, Ko YG, Yoon J, Lee C, Beom SH, Choi YD, Han WK, Ham WS, Han H, Lee J, Heo JE, Kim D, Baek ES, Kim S, Jung M, Shin SJ. Efficacy and Safety of Ifosfamide and Mesna in Metastatic Castration-Resistant Prostate Cancer after Taxane-Based Chemotherapy and Novel Hormonal Therapy Failure. Cancer Res Treat. 2025 Jun 9. doi: 10.4143/crt.2025.155. Online ahead of print. PMID 40506027